CLINICAL TRIAL: NCT04745169
Title: Home-Based Exercise as an Intervention to Treat Decreased Physical Function in Patients With Varying Levels of Kidney Function
Brief Title: Home-Based Exercise to Treat Decreased Physical Function in Patients With Varying Levels of Kidney Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Mayo Clinic (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Elizabeth Coite Lorenz, Principal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-52019
Record Dates: First submitted 2021-01-29; First posted 2021-02-09 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: This is a pilot study to be conducted at Baylor College of Medicine in Houston, TX examining the feasibility, safety, acceptability, and preliminary efficacy of home-based exercise on frailty parameters and SPPB score in patients with varying levels of kidney function. The effects of exercise on HRQOL, physical activity, and adverse outcomes including hospitalizations, will also be explored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Participants will be asked to complete an 8-week home-based exercise intervention
  Interventions: Behavioral: 8 week home-based exercise program

INTERVENTIONS:
Behavioral: 8 week home-based exercise program — Participants will be asked to complete an 8-week home-based exercise program according to guidelines from the American Heart Association and the American Association of Cardiovascular and Pulmonary Rehabilitation. At study baseline, participants will receive exercise equipment and an individualized exercise prescription from an exercise physiologist followed by 8 weekly phone calls from an exercise physiologist. Participant safety will be monitored.

SUMMARY:
The investigators will conduct a pilot study to determine whether home-based exercise is an effective intervention to improve decreased physical function in kidney transplant candidates. The investigators will determine if home-based exercise improves frailty parameters and SPPB scores. The investigators will also determine if home-based exercise improves health-related quality of life (HRQOL), physical activity, and adverse clinical outcomes, including hospitalizations.

DETAILED DESCRIPTION:
Screening and Recruitment:

Potential participants will be identified from dialysis units, nephrology clinics, primary care clinics, or kidney transplant clinics at Baylor College of Medicine. Patients who express interest in the study will go through the informed consent process with a member of the study team, and patients wishing to participate in the study will complete written consent. If patients have not had frailty and SPPB testing within the two weeks prior to consent, the study team member will perform frailty and SPPB testing at baseline in a supervised setting. Patients who are not frail or pre-frail and have a SPPB score > 10 will be ineligible for study participation.

Exercise Intervention:

Participants will be provided with a pedal exerciser, resistance bands, and exercise pamphlets. Participants will be asked to complete an 8-week home-based exercise program with a focus on the core components of physical activity counseling and exercise training according to guidelines from the American Heart Association and the American Association of Cardiovascular and Pulmonary Rehabilitation. Participants will receive an individualized exercise prescription. Recommended aerobic exercises will include arm and/or leg ergometry using a pedal exerciser, and recommended resistance training will include resistance bands. During the program, participants will receive weekly semi-scripted phone calls from an exercise physiologist and gradual increases in the volume of physical activity will be recommended over time. Participants will be asked to log information regarding their exercise sessions.

Study Measures:

Participants will complete the Short Physical Performance Battery (SPPB), and Fried Frailty phenotype at baseline and after completion of the exercise intervention. The SPPB consists of gait speed, balance, and repeat chair stand tests. The Fried Frailty Phenotype consists of gait speed and grip strength tests, in addition to self-reported measurement of physical activity, weight loss, and exhaustion. Participants will also be asked to complete questionnaires and wear a physical activity monitor at baseline and after completion of the exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Consenting to research
* Chronic kidney disease (stages 1-5)
* An SPPB score ≤10 or considered frail or pre-frail according to the Fried Frailty Phenotype

Exclusion Criteria:

* Younger than 18 years
* Patients being evaluated for combined organ transplantation
* Significant comorbidities that limit rehabilitation potential including pulmonary disease requiring continuous oxygen supplementation, active angina, critical aortic sclerosis, decompensated heart failure, or known ventricular arrhythmia.
* An SPPB score >10 or not considered frail or pre-frail by the Fried Frailty Phenotype
* Non-English speaker without availability of adequate interpreter services (safety concern)
* Failure to pass submaximal exercise test in patients not approved for kidney transplantation at our center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Lorenz, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 15
Completed | 9
Not Completed | 6
Not completed — Kidney transplantation | 1
Not completed — Participant health problems | 3
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [58 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White race | 11
Region of Enrollment [Number; unit: participants]
  United States | 15
Dialysis dependent [Count of Participants; unit: Participants] | 8
Diabetes [Count of Participants; unit: Participants] | 12
Never smoked [Count of Participants; unit: Participants] | 10
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 30.3 [27.7 to 37.6]
Physical Frailty Phenotype score [Median (Inter-Quartile Range); unit: units on a scale] — The Physical Frailty Phenotype score is based on 5 criteria: unintentional weight loss, exhaustion, low physical activity, slowness, weakness. Participants receive a score of 1 for each criterion they meet. The criterion scores are then summed to provide a total score ranging from 0-5 with higher scores indicating greater frailty. Specifically, a total score of 0 indicates that the participant is not frail, a score of 1-2 indicates that the participant is pre-frail, and a score of 3-5 indicates that the participant is frail.
  units on a scale | 2 [1 to 2]
Short Physical Performance Battery score [Median (Inter-Quartile Range); unit: units on a scale] — The Short Physical Performance Battery is a composite measure which includes component tests of balance, gait speed, and chair stand time. Participants receive a score of 0-4 for each of the 3 component tests with lower scores indicating worse physical function. Component scores are then summed providing a total score of 0-12 with lower scores again indicating worse physical function.
  units on a scale | 9 [8 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Change in Short Physical Performance Battery Score
Description: The Short Physical Performance Battery is a composite measure which includes component tests of balance, gait speed, and chair stand time. Participants receive a score of 0-4 for each of the 3 component tests with lower scores indicating worse physical function. Component scores are then summed providing a total score of 0-12 with lower scores again indicating worse physical function.
Time Frame: 8 weeks of home-based exercise
Population: Median difference in 8-week score compared to baseline score
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 9
units on a scale | -1 [-2 to 1.5]
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p = 0.73, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Grip Strength
Description: Grip strength will be measured using a hand-held dynamometer.
Time Frame: 8 weeks
Population: Median difference in 8-week grip strength compared to baseline
Measure: Median (Inter-Quartile Range); unit: kilograms
Arm/Group | Intervention
Number analyzed (Participants) | 9
kilograms | 2.8 [0.2 to 6.3]
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Gait Speed
Description: Gait speed at the participant's self-selected walking speed will be measured.
Time Frame: 8 weeks
Population: Median difference in 8-week gait speed compared to baseline
Measure: Median (Inter-Quartile Range); unit: meters/second
Arm/Group | Intervention
Number analyzed (Participants) | 9
meters/second | -0.1 [-0.3 to 0.2]
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p = 0.65, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Exhaustion
Description: Patients will self-report their level of exhaustion using the Center for Epidemiologic Studies Depression Scale (CES-D) which consists of a 4-point scale. Items on the CES-D are scored from minimum to maximum values (1 point to 4 points) which are indicated on the CES-D as "rarely or none of the time," "some or a little of the time," "occasionally or a moderate amount of time," "most or all of the time," respectively. A higher number of points indicates a worse outcome. Energy/fatigue scores on the Kidney Disease Quality of Life Short Form (KDQOL-SF) will also be calculated. Energy/fatigue scores range from 0 to 100 points with a higher number of points indicating a worse outcome.
Time Frame: 8 weeks
Population: Median difference in 8-week energy/fatigue score compared to baseline score
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 9
score on a scale | 10.0 [-5.0 to 20.0]
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Physical Activity
Description: Energy expenditure will be measured using an activity monitor worn on the wrist for 7 days. Low activity is defined as activity in the lowest 20% (<383 Kcals/week for men or <270 Kcals/week for women). Patients will also self-report their activity level using the Minnesota Leisure Time Physical Activity Questionnaire.
Time Frame: 8 weeks
Population: Median difference in moderate to vigorous physical activity at 8-week score compared to baseline
Measure: Median (Inter-Quartile Range); unit: hours per day
Arm/Group | Intervention
Number analyzed (Participants) | 9
hours per day | -0.4 [-1.3 to 0.4]
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p = 0.55, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Quality of Life
Description: Health-related quality of life will be measured using the Kidney Disease Quality of Life Short Form. This questionnaire includes scales with minimum values of 0 and maximum values of 100. Higher scores indicate better quality of life.
Time Frame: 8 weeks
Population: Median difference in 8-week mental health score compared to baseline score
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 8
score on a scale | 1.7 [-9.4 to 8.4]
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in Weight
Description: Weight will be measured using a scale.
Time Frame: 8 weeks
Population: Median difference in 8-week weight compared to baseline
Measure: Median (Inter-Quartile Range); unit: kilograms
Arm/Group | Intervention
Number analyzed (Participants) | 9
kilograms | -1.1 [-2.1 to 0.2]
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change in Percent Body Fat
Description: Change in percent body fat from baseline to 8 weeks was measured in the subset of participants from Mayo Clinic using bioelectrical impedance analysis.
Time Frame: 8 weeks
Population: Median difference in 8-week percent body fat compared to baseline
Measure: Median (Inter-Quartile Range); unit: percentage of body fat
Arm/Group | Intervention
Number analyzed (Participants) | 7
percentage of body fat | 0.9 [0 to 1.3]
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Physical Frailty Phenotype
Description: The Physical Frailty Phenotype score is based on 5 criteria: unintentional weight loss, exhaustion, low physical activity, slowness, weakness. Participants receive a score of 1 for each criterion they meet. The criterion scores are then summed to provide a total score ranging from 0-5 with higher scores indicating greater frailty. Specifically, a total score of 0 indicates that the participant is not frail, a score of 1-2 indicates that the participant is pre-frail, and a score of 3-5 indicates that the participant is frail.
Time Frame: 8 weeks
Population: Median difference in 8-week score compared to baseline score
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 9
units on a scale | 0 [-1 to 0]
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 3/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=15)
Transient musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Persistent musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT04745169/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT04745169/ICF_001.pdf